CLINICAL TRIAL: NCT04513249
Title: Effects of Therapeutic Plasmaexhange on Viscoelastic Tests in Non-coagulopathic Patients
Status: Completed | Type: Observational
Sponsor: Institutul Clinic Fundeni (Other)
Responsible Party: Principal Investigator, Popescu Mihai, Clinical Professor, Institutul Clinic Fundeni
Other Study IDs: FFP
Record Dates: First submitted 2020-08-11; First posted 2020-08-14 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Transfusion Related Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: dynamics of coagulation parameters — the effects of fresh frozen plasma administered during a plasma exchange therapy on viscoelastic tests

SUMMARY:
Therapeutic plasma exchange is widely performed in patients with autoimmune disease. The exact effects of fresh frozen plasma on coagulation in this group of patients remains unknown. In order to investigate this issue the present study monitors periprocedural coagulation status with the aid of standard coagulation tests and rotational thromboelastometry. Four thromboelastometric tests will be performed: ExTEM, InTEM, FibTEM and ApTEM. The following parameters will be recorded from each test: CT (sec), CFT (sec) and MCF (mm) one hour before and one hour after plasmaechange was performed.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing therapeutic plasma exchange for autoimmune disease

Exclusion Criteria:

* previous coagulation disorders
* anticoagulant or antiplatelet therapy within the last 7 days

Min Age: 18 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: consecutive patients undergoing therapeutic plasmaechange for autoimmune disease
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
change in clotting time - CT (%) | one hour before compared to one hour after plasmaexchange
  change in CT determined before and after plasmaexchange. A 20% change in parameter value will be considered clinically significant.

SECONDARY OUTCOMES:
change clot formation time - CFT (%) | one hour before compared to one hour after plasmaexchange
  change in CFT determined before and after plasmaexchange. A 20% change in parameter value will be considered clinically significant.
change maximum clot firmness - MCF (%) | one hour before compared to one hour after plasmaexchange
  change in MCF determined before and after plasmaexchange. A 20% change in parameter value will be considered clinically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Dana Tomescu, Prof, Study Chair — Fundeni Clinical Institute
Locations (1):
- Fundeni Clinical Institute, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No